CLINICAL TRIAL: NCT01323985
Title: A Phase 1 Dose Escalation Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Single Intravenous Doses of GSK2315698A in Healthy Volunteers
Brief Title: SAP Depleter Dose Escalation Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113776
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — miridesap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2315698 (Experimental): Intravenous infusion single dose
  Interventions: Drug: GSK2315698

INTERVENTIONS:
Drug: GSK2315698 — 5mg-400mg IV (in the vein) single dose over 1-4 hours
Drug: GSK2315698 — IV (in the vein) single dose over 24 hours, in two sessions

SUMMARY:
The purpose of this study is to provide safety information and to define the optimal induction and short term maintenance regimen for GSK2315698 to deplete circulating SAP in healthy volunteers prior to assessing in patients

DETAILED DESCRIPTION:
This single centre, open label, dose escalation study is designed to assess safety (including adverse events, vital signs, ECGs, and clinical laboratory tests), and pharmacokinetic /pharmacodynamic parameters in healthy volunteers. Subjects will attend for 3 sessions: session 1 is a single intravenous (IV) infusion over a short time period to confirm the safety of a single dose of GSK2315698 over a wide dose range, sessions 2 and 3 will investigate IV infusion regimens over 24 hours (induction phase followed by maintenance phase). The dosing regimen will be adjusted adaptively to optimise the induction and maintenance phases of the dosing regimen. amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. (As a precaution a pregnancy test will be conducted prior to dosing; a positive test will lead to exclusion).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol Section 8.1. This criterion must be followed from the time of the first dose of study medication until 85 days post-last dose.
* Body weight gretaer than or equal to 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTc, < 450 msec
* Peripheral veins suitable for venous blood sampling and cannulation
* Smokers (<10 /day) are permitted but must be willing to abstain for the duration of residential study sessions

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Previous surgical procedures on the upper digestive tract including cholecystectomy (gallbladder removal), and/or cholelithotomy (gallstone removal).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 84 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01-06 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
An assessment of the safety and tolerability of single intravenous dose of GSK2315698 | 12 weeks
To characterize the PK/PD relationship GSK2315698 in order to define an intravenous dosing regimen that provides optimal depletion of blood SAP over a 24 hour period (in healthy volunteers) | 12 weeks

SECONDARY OUTCOMES:
Measure the pharmacokinetics of IV administration of GSK2315698 | 12 weeks
Measure depletion of SAP following IV administration of GSK2315698 | 12 weeks
Measure the kinetics of SAP production and SAP degradation in healthy volunteers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 113776 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113776?search=study&study_ids=113776#rs